CLINICAL TRIAL: NCT01373879
Title: Safety and Immunogenicity of Heterologous Prime-boost With the Candidate Malaria Vaccines AdCh63 ME-TRAP and MVA ME-TRAP in Healthy Adults and Children in a Malaria Endemic Area
Brief Title: AdCh63 ME-TRAP and MVA ME-TRAP Malaria Vaccines Evaluation in Healthy Adults and Children in a Malaria Endemic Area
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC041
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Malaria
Keywords: Vaccine; Immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1A (Experimental): Adults (18-50 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 1B (Experimental): Adults (18-50 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 2A (Experimental): Children (2-6 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 2B (Experimental): Children (2-6 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 2C (Active Comparator): Children (2-6 years old) vaccinated with human diploid cell rabies vaccine
  Interventions: Biological: HDCRV
- Group 3A (Experimental): Children (2-6 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 3B (Experimental): Children (2-6 years old) vaccinated with AdCh63 ME-TRAP followed with MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group 3C (Active Comparator): Children (2-6 years old) vaccinated with human diploid cell rabies vaccine
  Interventions: Biological: HDCRV

INTERVENTIONS:
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 1 x 10^10vp IM followed by MVA ME-TRAP 2 x 10^8 pfu IM 8 weeks later
  Arms: Group 1A
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 5 x 10^10vp IM followed by MVA ME-TRAP 2 x 10^8 pfu IM 8 weeks later
  Arms: Group 1B
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 1 x 10^10vp IM followed by MVA ME-TRAP 1 x 10^8 pfu IM 8 weeks later
  Arms: Group 2A
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 1 x 10^10vp IM followed by MVA ME-TRAP 2 x 10^8 pfu IM 8 weeks later
  Arms: Group 2B
Biological: HDCRV — HDCRV 1ml IM followed by HDCRV 1ml IM 8 weeks later
  Arms: Group 2C
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 5 x 10^10vp IM followed by MVA ME-TRAP 1 x 10^8 pfu IM 8 weeks later
  Arms: Group 3A
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — AdCh63 ME-TRAP 5 x 10^10vp IM followed by MVA ME-TRAP 2 x 10^8 pfu IM 8 weeks later
  Arms: Group 3B
Biological: HDCRV — HDCRV 1ml IM followed by HDCRV 1ml IM 8 weeks later
  Arms: Group 3C

SUMMARY:
The purpose of this trial is to assess the safety and immunogenicity of MVA ME-TRAP and AdCH63 ME-TRAP candidate vaccines in healthy children and adult volunteers in a malaria endemic region. The regimen proposed here has protected non-immune volunteers in Oxford against sporozoite challenge, and so may be protective against naturally acquired infection in The Gambia.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult males aged 18-50 years in good health and healthy children aged 2-6 years.with consenting parents.

Exclusion Criteria:

* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
* Severe malnutrition.
* Hypersensitivity to HDCRV.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, betapropiolactone.
* History of splenectomy Haemoglobin less than 9.0 g/dL, where judged to be clinically significant in the opinion of the investigator
* Serum Creatinine concentration greater than 70 mol/L, where judged to be clinically significant in the opinion of the investigator
* Serum ALT concentration greater than 45 U/L, where judged to be clinically significant in the opinion of the investigator
* Blood transfusion within one month of enrolment.
* History of vaccination with previous experimental malaria vaccines.
* Administration of any other vaccine or immunoglobulin within two weeks before vaccination.
* Current participation in another clinical trial, or within 12 weeks of this study.
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area.
* HIV positive.
* Positive malaria antigen test

Ages: 2 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety of a heterologous prime-boost vaccine strategy with AdCh63 ME-TRAP and MVA ME-TRAP | Participants will be followed for the duration of the study, an expected average of 12 months
  To assess the safety of a heterologous prime-boost vaccine strategy with AdCh63 ME-TRAP and MVA ME-TRAP in healthy adults and children in The Gambia by recording local and systemic solicited and unsolicited adverse events

SECONDARY OUTCOMES:
Immunogenicity of a heterologous prime-boost vaccine strategy with AdCh63 ME-TRAP and MVA ME-TRAP | Participants will be followed for the duration of the study, an expected average of 12 months
  To assess the immunogenicity of a heterologous prime-boost vaccine strategy with AdCh63 ME-TRAP and MVA ME-TRAP in healthy adults and children in The Gambia by assessing induced antibody and T cell response to the vaccine insert.

CONTACTS AND LOCATIONS:
Overall Officials: Kalifa Bojang, Principal Investigator — Medical Research Council PO Box 273, Banjul The Gambia
Locations (1):
- Dr Kalifa Bojang, Banjul, The Gambia

REFERENCES:
- [Derived] Ogwang C, Afolabi M, Kimani D, Jagne YJ, Sheehy SH, Bliss CM, Duncan CJ, Collins KA, Garcia Knight MA, Kimani E, Anagnostou NA, Berrie E, Moyle S, Gilbert SC, Spencer AJ, Soipei P, Mueller J, Okebe J, Colloca S, Cortese R, Viebig NK, Roberts R, Gantlett K, Lawrie AM, Nicosia A, Imoukhuede EB, Bejon P, Urban BC, Flanagan KL, Ewer KJ, Chilengi R, Hill AV, Bojang K. Safety and immunogenicity of heterologous prime-boost immunisation with Plasmodium falciparum malaria candidate vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, in healthy Gambian and Kenyan adults. PLoS One. 2013;8(3):e57726. doi: 10.1371/journal.pone.0057726. Epub 2013 Mar 19. PMID 23526949